CLINICAL TRIAL: NCT04520984
Title: A Pilot Randomized-Controlled Study Of The Impact Of Integrated Palliative And Nephrology Care Versus Usual Nephrology Care On Symptom Burden, Quality Of Life And Advance Care Planning In Patients With Chronic Kidney Disease Stage V Not On Dialysis
Brief Title: Pilot Randomized-controlled Trial of Integrated Palliative and Nephrology Care Versus Usual Nephrology Care.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-01259
Record Dates: First submitted 2020-08-18; First posted 2020-08-20 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Intervention
  Interventions: Other: Integrated ambulatory palliative and nephrology care
- Arm 2 (Other): Standard Care
  Interventions: Other: Standard nephrology care

INTERVENTIONS:
Other: Integrated ambulatory palliative and nephrology care — Monthly ambulatory care visits with the kidney palliative care team in the intervention group for three months.
  The intervention in this study is addition of a palliative care team to the care team of the subject. This intervention will not change or impact their regular nephrology care. The subjects in the intervention arm will be seen by the palliative care team three times over the 12-week study period (once per month).The intervention will be delivered by a physician trained in both palliative care and nephrology, the PI of the study.
  Arms: Arm 1
Other: Standard nephrology care — Standard nephrology care
  Arms: Arm 2

SUMMARY:
The objective of this application is to conduct a pilot study testing the impact of integrated nephrology and palliative care versus standard nephrology care on patient-reported outcomes. This study is a preliminary study designed to determine feasibility of a palliative care study inclusive of kidney disease patients and to look for trends in impact over a 12-week follow-up period. Measurements will be taken at time one (time of enrollment) and time two (12 weeks). Our central hypothesis is that integration of palliative care with standard nephrology care in the ambulatory care of patients with a glomerular filtration rate (eGFR) ≤15ml/min/1.73m2 will trend towards improved symptom control, quality of life, and increased documentation of advance care planning when compared to usual nephrology care. We expect 10-15 patients per arm.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Age ≥18
2. Fluent English speaker
3. eGFR≤15 mL/min/1.73m2 (diagnosis of CKD stage V)
4. Able to give consent
5. Must be followed by a faculty group practice nephrologist

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Diagnosis of dementia
2. Non-English speaker
3. Have been seen by a palliative care provider prior to study entry
4. Pregnant women
5. On dialysis or have received a kidney transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-07-12 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Change in IPOS-Renal symptom assessment score | Baseline, week 12
  IPOS-Renal is a short measure (11 questions), combining the most common symptoms renal patients experience plus additional items from IPOS on concerns beyond symptoms, such as information needs, practical issues, family anxiety. The total score reflects symptom burden and can range from zero to 68, where 0 is least symptom burden and 68 is highest symptom burden.
Change in KDQOL-SF 36 Quality of Life Scores | Baseline, week 12
  The KDQOL-36 has five scales, including two generic HRQOL scales from the SF-12 version 1 (12 items total) and three kidney-specific scales (24 items total). The SF-12 PCS and MCS are scored on a T-score metric (mean=50, SD=10, in the United States general population), with higher scores indicating better HRQOL.
Difference between the number of documented advanced care planning between arms | Week 12
  advanced care planning = health care proxy, Medical Order for Life Sustaining Treatment [MOLST], or a Do Not Resituate form

SECONDARY OUTCOMES:
retention patients at the end of the study | 12 weeks
percent of returned clinical surveys (IPOS-R and KDQOL-SF 36 | 12 weeks
patient satisfaction as rated on the Press Ganey Survey | 12 weeks
  Measure satisfaction on a five point scale where "5" is the Top Score.

OTHER OUTCOMES:
Change in IPOS-Renal symptom assessment score over time in intervention arm | Baseline, 6 weeks, 12 weeks
  Exploratory end-points include change in symptom burden over time in the intervention arm. These subjects are expected to have three visits with symptom surveys filled out at each visit. We hypothesize that symptom burden will improve over time.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Scherer, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to the PI. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Scherer JS, Rau ME, Krieger A, Xia Y, Zhong H, Brody A, Charytan DM, Chodosh J. A Pilot Randomized Controlled Trial of Integrated Palliative Care and Nephrology Care. Kidney360. 2022 Aug 12;3(10):1720-1729. doi: 10.34067/KID.0000352022. eCollection 2022 Oct 27. PMID 36514730